CLINICAL TRIAL: NCT00601679
Title: Improvement in Clinical Outcomes of Patients With Chronic Heart Failure Using Serial NT-proBNP Monitoring: The EX-IMPROVE-CHF Study
Brief Title: Improvement of Patients With Chronic Heart Failure Using NT-proBNP
Acronym: EXIMPROVECHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN0013
Record Dates: First submitted 2008-01-08; First posted 2008-01-28 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Congestive Heart Failure
Keywords: CHF treatment&prognosis,NT-proBNP testing.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NT-proBNP (Experimental): Surveillance NT-proBNP levels disclosed to physicians. Intervention (e.g. Diuretic management) based on NT-proBNP results.
  Interventions: Other: NT-proBNP guided care
- Usual Care (No Intervention): Surveillance NT-proBNP levels blinded. Intervention (e.g. Diuretic management) based on clinical judgments.

INTERVENTIONS:
Other: NT-proBNP guided care — knowledge of NT-proBNP results
  Arms: NT-proBNP

SUMMARY:
This will be a multicentre Phase IV study in which patients with chronic HF who are managed and followed by HF/heart functions clinics will be followed over a period of two years.

Clinic patients who are recruited into the study will have obligatory blood sampling for the surveillance measurement of NT-proBNP level every three months for a minimum of one year (4 samples). One-half of the subjects in each clinic will be randomized to have these NT-proBNP values made known to the attending clinic physicians and nurses, the other half will have these values blinded. During the study, attending clinic physicians can order open-label NT-proBNP or BNP assays, if available in their institution, to assist the management of their patients if they feel it is clinically needed.

DETAILED DESCRIPTION:
Once an eligible clinic patient is identified, written informed consent will be obtained. All patients will have blood drawn for the measurement of NT-proBNP immediately after consent is obtained. The patient will then be randomized to either the usual care or NT-proBNP arm.

For each patient enrolled into the study the attending physician will ensure obligatory blood sampling for the measurement of NT-proBNP level every three months for a minimum of one year (4 samples). Conventional measures used in programmed management settings including history taking, physical and radiographic examination and echocardiography will also be undertaken as per clinical practice. Patients from both arms will be treated with the same conventional measures.

One-half of the subjects in each clinic will be randomized to have these NT-proBNP values made known to the attending clinic physicians and nurse practitioners. The other half (Usual Care) will have these values blinded. During the study, attending clinic physicians can order NT-proBNP or BNP assays, if available in their institution, to assist the management of their patients if they feel it is clinically needed. Demographic variables such as age, gender, BMI, serum creatinine, and eGFR will also be collected in both arms. A dedicated research coordinator based in St. Michael's Hospital, the core centre, will monitor patients, data and blood sample collection from all participating clinics. NT-proBNP will be measured on site in clinics with the facility to measure NT-proBNP. For clinics that do not have the facility, the samples will be shipped to the core centre for measurement and the results will be provided to the clinic within one week for those patients who are randomized to open-label NT-proBNP. The research coordinator, via close communications with the clinic nurses and physicians, will ensure the process is immaculately executed and blinding is maintained.

All patients will be followed every three months for a minimum of one year (4 samples) and will include an initial evaluation (Visit 1) along with four follow-up visits in the HF/heart functions clinics (Visits 2 - 5). A clinic visit will be requested for those patients having experienced a serious adverse event since Visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* NYHA class II-IV heart failure
* Followed in a programmed heart failure (HF) management setting

Exclusion Criteria:

* Life expectancy <1 year due to causes other than HF such as advanced cancer
* Any other conditions that may render the patient ineligible according to the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Heart failure hospitalization and death | 2 years

SECONDARY OUTCOMES:
Time to hospitalization/admission to ED due to HF, total number of HF events, total number of hospitalizations for cardiovascular events, all-cause mortality, cardiovascular mortality, worsening in clinical status but not requiring hospital admission | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W Moe, MD, FACC, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St Michael's Hospital, Toronto, Ontario